CLINICAL TRIAL: NCT00175630
Title: Effect of Femoral Nerve Block on Opioid Requirements Following Anterior Cruciate Ligament Reconstruction: A Double Blind, Prospective Randomized Controlled Trial
Brief Title: The Effect of Femoral Nerve Block on Postoperative Opioid Use After Anterior Cruciate Ligament (ACL) Reconstruction
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H05-70078; W05-0024
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Pain, Postoperative
Keywords: ACL reconstruction; morphine sparing; preemptive analgesia; Post-operative pain and post- operative opioid use
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Administration of a femoral nerve block (bupivacaine HCL) — See Detailed Description

SUMMARY:
This study evaluates the effect of a femoral nerve block on opioid requirements following anterior cruciate ligament (ACL) reconstruction. This is a double blind, prospective randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Schedule for primary elective anterior cruciate ligament reconstruction
* Tolerance to bupivacaine
* Tolerance to non-steroidal anti-inflammatory drugs (NSAIDs)
* Informed consent

Exclusion Criteria:

* Patients who received a femoral nerve block more than 1 hour prior to surgery
* Complex associated injuries or pre-existing conditions that will delay time to ambulation
* Children with tibial avulsion fractures
* Allergic and/or sensitive to bupivacaine and/or NSAIDs
* 30% over ideal body weight
* Acute ACL reconstruction (done less than 2 weeks after injury)
* Pre-existing femoral nerve injury
* Psychiatric patients on psychotropic agents
* History of drug or alcohol dependence or recreational drug use
* Refusal to provide informed consent

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative morphine requirement

SECONDARY OUTCOMES:
Pain rating | immediately post-op
Opioid surgical time | time from end of anaesthesia to first requirement of morphine

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Reilly, MD, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Department of Orthopaedics, Vancouver, British Columbia, Canada